CLINICAL TRIAL: NCT03679910
Title: Evaluation of Cell Migration Inducing Protein (CEMIP) in Diagnosis of Pancreatic Carcinoma in Comparison With Other Traditional Markers
Brief Title: Evaluation of CEMIP in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Safwat, doctor, Assiut University
Other Study IDs: CEMIP in pancreatic cancer
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Pancreas Cancer
Keywords: CA 19-9; CEA
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Liver Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: pancreatic cancer patients (50 patients)
  Interventions: Diagnostic Test: CEMIP , CA19-9 ,CEA; Diagnostic Test: A) CBC . B) RBG. C)KFT. D) LFT.
- Group2: A- Non-pancreatic cancer subjects with benign diseases will be 20 subjects. B- Healthy individuals (control): 20 apparently healthy volunteers after informed consent.
  Interventions: Diagnostic Test: CEMIP , CA19-9 ,CEA; Diagnostic Test: A) CBC . B) RBG. C)KFT. D) LFT.

INTERVENTIONS:
Diagnostic Test: CEMIP , CA19-9 ,CEA — CEMIP: Cell migration inducing protein CA19-9: Carbohydrate antigen 19-9 CEA: Carcinoembryonic antigen
Diagnostic Test: A) CBC . B) RBG. C)KFT. D) LFT. — A)CBC: Complete blood count. B)RBG: Random blood glucose. C)KFT: Kidney function tests. D)LFT: Liver function tests.

SUMMARY:
Pancreatic cancer (PC) is one of the most lethal diseases among all cancer types.

The diagnosis of PC is usually based on radiology or invasive endoscopic techniques. Various types of tumor markers are used for diagnosing PC. The tumor markers carbohydrate antigen19-9 (CA 19-9) and carcinoembryonic antigen (CEA) are the ones most closely tied to PC. These tests are more often used in people already diagnosed with pancreatic cancer to help tell if treatment is working or if the cancer is progressing .

Cell migration inducing protein (CEMIP) has been reported to be associated with early detection, cancer cell migration, invasion, and poor prognosis.

Aim of the work:

* To Estimate the level of CEMIP, CA19-9 and CEA in pancreatic cancer patients.
* To evaluate the clinical utility of serum CEMIP, CA19-9 and CEA in pancreatic cancer patients in comparison with healthy controls and their relation to cancer staging and histopathological types.
* To detect the correlation between CEMIP, CA-19-9 and CEA.

DETAILED DESCRIPTION:
Pancreas is an important retroperitoneal organ with exocrine and endocrine functions. Pancreatic cancer (PC) is one of the most lethal diseases among all cancer types. It moved from the fourth to the third leading cause of cancer-related death in the United States and is anticipated to become the second around 2020. It accounts for about 3% of all cancers in the United State and about 7% of all cancer deaths.

The estimated number of PC cases in Egypt in 2013 was 2,226, and it is projected to increase and be 2,836 and 6,883 in 2020 and 2050 respectively. The overall age-adjusted PC mortality rate in Egypt was 1.47/100,000 population and analysis of the regional distribution showed significant variations in rates among provinces with Northern provinces having higher rates than Southern regions.

The asymptomatic nature of early PC, the lack of sensitive and specific tools to diagnose early disease, and the lack of response to most forms of treatment all contribute to the high mortality rate of pancreatic cancer. This poor outcome could be largely due to the late diagnosis. The expression profiles of PC had been widely studied, revealing several molecular factors affecting various aspects of PC.

Tumors of pancreas are divided into: Non-endocrine tumors which maybe benign or malignant and endocrine tumors.

The diagnosis of PC is usually based on radiology [computed tomography (CT) and magnetic resonance imaging (MRI)] or invasive endoscopic techniques [ultrasound endoscopy-fine needle aspiration (EUS-FNA), endoscopic retrograde cholangiopancreatography (ERCP), and explorative laparoscopy. Imaging diagnosis method is a normal method for clinical tumor diagnosis. But due to the various defects of the image device, it is usually to combine several kinds of technologies for diagnosis. Moreover because of the low sensitivity and specificity, the methods are often used in the diagnosis of high risk groups, rather than early detection. Therefore, it is urgently needed to develop new methods for early diagnosis of cancer.

An ideal diagnostic method for PC should definitively distinguish malignant lesions from benign lesions, provide precise tumor staging, and detect early-stage disease and preneo-plastic conditions. There are many challenges in the early detection of PC, including its asymptomatic nature, the lack of a characteristic radiological manifestation and the absence of specific molecules in body fluid. Therefore, convenient and highly sensitive diagnostic tests for screening PC are probably more important than tests with good specificity but moderate sensitivity.

Various types of tumor markers are used for diagnosing PC. The tumor markers carbohydrate antigen19-9(CA 19-9) and carcinoembryonic antigen (CEA) are the ones most closely tied toPC. But these proteins don't always go up when a person has pancreatic cancer, and even if they do, the cancer is often already advanced by the time this happens. Sometimes levels of these tumor markers can go up even when a person doesn't have pancreatic cancer. For these reasons, CA19-9 and CEA aren't used to screen for pancreatic cancer, although a doctor might still order these tests if a person has symptoms that might be from pancreatic cancer. These tests are more often used in people already diagnosed with pancreatic cancer to help tell if treatment is working or if the cancer is progressing.

Although CA 19-9 is known as a pancreatic cancer biomarker, it is not commonly used for general screening, owing to its low sensitivity and specificity. In particular, false-negative results in the segment of the population with Lewis blood type A-B- and false-positive results in patients with obstructive jaundice limit the specificity of CA 19-9 for PC. Therefore, development of novel diagnostic markers is required for the early detection of PC.

CEMIP (KIAA1199), defined as cell migration inducing protein currently is located in chromosome 15q25.1, which appears in the nucleus and cytoplasm. It is a secreted protein (153KDa) rather than a transmembrane protein. Its mutation site was reported to cause hearing loss due to the folding change of protein structure, meanwhile the over-expression of CEMIP referred to dreadful invasion and uncontrolled proliferation of tumor with distant metastasis and limited survival opportunity of patients. Especially, over-expressed CEMIP also protected malignant tumor from strict microenvironment in hypoxia, low glucose and cracked barrier, leading to enhanced adaptability of tumor by stimulating the epidermal growth factor receptor (EGFR), fibroblast growth factor receptors (FGFR) pathway. CEMIP plays an important role in cytokine pathway and its over-expression in tumors provide a novel target for individual therapy. Targeting CEMIP would thereby dysregulate the cytokine pathway which would in turn, decide the growth and death of the vicious tumor cells.

Increased expression of CEMIP has been reported in various cancers including: breast, colorectal and gastric. Several studies have investigated the role of CEMIP in pancreatic cancer. It has been reported to be associated with early detection, cancer cell migration, invasion, and poor prognosis. Suh., 2016 suggested that CEMIP may be useful for detecting pancreatic cancer at an early stage, while Koga., 2017 demonstrated its association with prognosis in PC.

Primary screening using circulating biomarkers followed by confir¬mative diagnosis based on imaging and patho¬logic results might be the future strategy for diagnosing PC.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

Includes all patients presented by pancreatic cancer with clinical, radiological, laboratory diagnosis and pathological diagnosis.

Group 2:

A: Healthy individual B: Individual with benign diseases such as benign hepatopancreatobiliary conditions as gall stones, obstructive calcular jaundice, chronic pancreatitis and benign gasrtrointestinal as ulcer and polyp.

Exclusion Criteria:

* Patients recently operated for pancreatic cancer.
* patients diagnosed to have another type of cancer (Breast, gastric or colorectal).
* High risk group of another type of cancer.
* Patients with disseminated cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on 90 informed individuals (according to the guidelines of ethical committee of faculty of Medicine, Assiut University and South Egypt Cancer Institute).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of cell migration inducing protein (CEMIP) in serum of pancreatic cancer as non invasive marker. | 2 day
  Measurement of CEMIP by enzyme linked immunosorbent assay (ELISA) in serum of pancreatic cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamel, MD, Principal Investigator — Assiut University; Omnia Abd El Monaem, MD, Study Chair — Assiut University; Randa Ahmed, MD, Study Chair — Assiut University; Dina Mohammed, Dr, Study Director — Assiut University
Locations (1):
- Dina Mohammed Safwat, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee HS, Jang CY, Kim SA, Park SB, Jung DE, Kim BO, Kim HY, Chung MJ, Park JY, Bang S, Park SW, Song SY. Combined use of CEMIP and CA 19-9 enhances diagnostic accuracy for pancreatic cancer. Sci Rep. 2018 Feb 21;8(1):3383. doi: 10.1038/s41598-018-21823-x. PMID 29467409
- [Background] Koga A, Sato N, Kohi S, Yabuki K, Cheng XB, Hisaoka M, Hirata K. KIAA1199/CEMIP/HYBID overexpression predicts poor prognosis in pancreatic ductal adenocarcinoma. Pancreatology. 2017 Jan-Feb;17(1):115-122. doi: 10.1016/j.pan.2016.12.007. Epub 2016 Dec 18. PMID 28012880
- [Background] Li L, Yan LH, Manoj S, Li Y, Lu L. Central Role of CEMIP in Tumorigenesis and Its Potential as Therapeutic Target. J Cancer. 2017 Jul 20;8(12):2238-2246. doi: 10.7150/jca.19295. eCollection 2017. PMID 28819426